CLINICAL TRIAL: NCT00794391
Title: Effects of a Brief Motivational Intervention on Risky Injection Practices Among Injecting Drug Users
Brief Title: Effects of Motivational Interviewing on Risky Injecting Practices Among Injecting Drug Users (IDUs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Karine Bertrand, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 13940 (FRSQ ID)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: HIV; Hepatitis C
Keywords: Vulnerable Populations; Injecting drug users; IDU; Risky injecting practices; Psychotherapy, brief; Motivational interviewing; Educational activities; Clinical trial; Risk behavior; risk reduction behavior
MeSH Terms: conditions — Hepatitis C; Risk-Taking; Risk Reduction Behavior | interventions — Motivational Interviewing; Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational interviewing (Experimental): Motivational interviewing is a client-centered, directive method for enhancing intrinsic motivation to change by exploring and resolving ambivalence (Miller & Rollnick. 1993). This 45 minutes individual motivational intervention focuses on risky injection practices.
  Interventions: Behavioral: Motivational interviewing
- Educational intervention (Active Comparator): The educational intervention is a 45 minutes individual intervention based on a document written by the Québec ministry of health (Québec, Canada). The aim is to inform participants about safe injection practices and to show them how to use sterile injection equipment.
  Interventions: Behavioral: Educational intervention

INTERVENTIONS:
Behavioral: Motivational interviewing — Motivational interviewing is a client-centered, directive method for enhancing intrinsic motivation to change by exploring and resolving ambivalence (Miller & Rollnick. 1993). This 45 minutes individual motivational intervention focuses on risky injection practices.
  Arms: Motivational interviewing
Behavioral: Educational intervention — The educational intervention is a 45 minutes individual intervention based on a document written by the Québec ministry of health (Québec, Canada). The aim is to inform participants about safe injection practices and to show them how to use sterile injection equipment.
  Arms: Educational intervention

SUMMARY:
The purpose of this study is to evaluate the effects of a brief motivational intervention in reducing risky injection practices among injecting drug users (IDUs). The investigators hypothesis is that motivational intervention will be more effective than educational intervention in reducing risky injection practices among IDUs.

DETAILED DESCRIPTION:
Injecting drug users (IDUs) are among the most vulnerable populations at risk to contract human immunodeficiency virus (HIV) and hepatitis C virus (HCV). Among Canadian cities, Montreal holds one of the higher HIV and HCV contraction rates in the IDU population. Results from SurvUDI, a population survey among IDUs conducted in the province of Quebec (Canada), show that in Montreal 18% of IDUs are infected with HIV and 67% are infected with HCV. The cornerstone of HIV and HCV prevention strategies is to give information on safe injection practices and to make available sterile syringes and other injection equipment. However, the SurvUDI survey reveals that a large proportion of IDUs recruited in community programs offering sterile injection equipment and information on safe injection practices are still sharing needles with other IDUs. Indeed, it seems that information dissemination and distribution of sterile injection equipment are not sufficient in order to control the HIV and HCV epidemic among IDUs. As a matter of fact, it is obvious that complementary interventions such as behavioural interventions are required. Motivational interviewing is an intervention technique centered on the individual. It aims to enhance intrinsic motivation to change behavior by helping the individual to resolve ambivalence. The scientific literature indicates that brief motivational intervention is a significantly effective intervention in order to reduce drug use problems and other related health problems. Furthermore, motivational intervention is well adapted for IDUs' resistance to change and their difficulties related with involvement in long-term therapeutic process. The present study's hypothesis is that IDUs assigned to the experimental group (brief motivational intervention) will present a greater diminution of their risky injection practices in comparison with IDUs assigned to the control group (educational intervention).

ELIGIBILITY:
Inclusion Criteria:

* In the last month, at least one cocaine injection
* In the last month, at least one injection with a syringe or another piece of injection equipment that has been used by someone else
* 16 years old or more
* French speaking
* Being able to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Risky injecting practices | 3 and 6 month follow-ups

SECONDARY OUTCOMES:
Stages of change for risky injecting practices (adapted from Prochaska & DiClemente) | 3 and 6 month follow-ups
Drug use (including injecting frequency) | 3 and 6 months follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Karine Bertrand, Ph.D., Principal Investigator — Université de Sherbrooke; Élise Roy, MD, MSc, Study Chair — Université de Sherbrooke; Carole Morissette, MD, FRCPC, Study Chair — Université de Montréal & Direction de santé publique de Montréal; Jean-François Boivin, MD, FRCPC, Study Chair — McGill University
Locations (1):
- Université de Sherbrooke, service de toxicomanie (Campus Longueuil), Montreal, Quebec, Canada